CLINICAL TRIAL: NCT03926104
Title: Evaluation of BNP Values in Major Vascular Surgery
Brief Title: BNP and Vascular Surgery
Acronym: BNPinVasc
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Clinical Professor, University of Parma
Other Study IDs: 39751 del 19/10/2018
Record Dates: First submitted 2019-01-07; First posted 2019-04-24 (Actual); Last update posted 2019-04-24 (Actual); Status verified 2019-04

CONDITIONS: General Anesthesia; Vascular Surgery; Abdominal Aortic Aneurysm; Natriuretic Peptide, Brain; Mets; Preoperative Period; Postoperative Period
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background and rationale of the study:

Patients undergoing non-cardiac major surgery show a perioperative cardiac risk and postoperative complications, that can be stratified based on parameters linked to patient's conditions and to surgery types.

An accurate identification of this risk could offer numerous advantages for these patients, who's 30-day mortality is around 2%. The identification of the correct risk could lead to a better pre- and postoperative management, that could guarantee a better surgery outcome and a faster postoperative recovery.

To this day there is no perfect method to correctly estimate this risk. Various studies show that high BNP levels are linked to cardiac events at 30 and 180 days. Further investigations identify different groups, at low, intermediate and high risk, based on BNP levels.

BNP is released by ventricular myocytes in response to a wall distress, due to an increased volume, pressure or myocardial ischemia.

So BNP plasma levels could be used as a prognostic and diagnostic marker, improving the cardiac risk stratification in patients undergoing surgery and a much more precise management.

This study is determined to do an evaluation of the correlations between pre- and postoperative BNP levels and the incidence of cardiac events in patients undergoing major vascular surgery.

DETAILED DESCRIPTION:
Patient's informed consent signature for adhesion at the study will be initially requested. With their acceptance, parameters will be recorded anonymously in the Case Report Form, identified by their initials and a numeric code, until hospital discharge.

The parameters analyzed will be related to:

* preoperative evaluation: anamnesis, health general conditions, METs, preoperative monitoring, in particularly BNP basal levels;
* intraoperative evaluation: intraoperative monitoring;
* postoperative evaluation: BNP and cTnI levels at 24 and 48 hours, and about pulmonary, cardiovascular, neurological and surgical postoperative complications, based on the medical record.

The data will be transferred on Excel worksheet, utilized for descriptive analysis related at every variable.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide an informed consent
* Age >18 years old
* Elective abdominal aortic aneurysm surgery

Exclusion Criteria:

* Emergency surgery
* Age ˂ 18 years old
* Creatinine >2mg/dl
* Diseases of ascending aorta, aortic arch or thoracic aorta
* Chronic atrial fibrillation
* Patient refusal to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult undergoing major vascular surgery
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2020-12-10 (Estimated); Study Completion 2020-12-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of cardiac events | from the induction of general anesthesia until hospital discharge, an average of 1 week

SECONDARY OUTCOMES:
Incidence of postoperative pulmonary complication | from immediately after surgery until hospital discharge, an average of 1 week
Incidence of postoperative neurological complication | from immediately after surgery until hospital discharge, an average of 1 week
Incidence of postoperative acute kidney failure | from immediately after surgery until hospital discharge, an average of 1 week
Incidence of unplanned ICU admission | from immediately after surgery until hospital discharge, an average of 1 week
Hospital length of stay | from immediately after surgery until hospital discharge, an average of 1 week
Incidence of mortality | from immediately after surgery until hospital discharge, an average of 1 week

CONTACTS AND LOCATIONS:
Locations (1):
- Elena Giovanna Bignami, Parma, Italy

REFERENCES:
- [Background] Vetrugno L, Orso D, Matellon C, Giaccalone M, Bove T, Bignami E. The Possible Use of Preoperative Natriuretic Peptides for Discriminating Low Versus Moderate-High Surgical Risk Patient. Semin Cardiothorac Vasc Anesth. 2018 Dec;22(4):395-402. doi: 10.1177/1089253217752061. Epub 2018 Jan 13. PMID 29332544
- [Background] Wayne Causey M, Singh N. Clinical implications of B-type natriuretic peptide and N-terminal pro--B-type natriuretic peptide in the care of the vascular surgery patient. Semin Vasc Surg. 2014 Dec;27(3-4):143-7. doi: 10.1053/j.semvascsurg.2015.01.004. Epub 2015 Jan 21. PMID 26073822
- [Background] Biccard BM, Devereaux PJ, Rodseth RN. Cardiac biomarkers in the prediction of risk in the non-cardiac surgery setting. Anaesthesia. 2014 May;69(5):484-93. doi: 10.1111/anae.12635. PMID 24738805
- [Background] Bryce GJ, Payne CJ, Gibson SC, Byrne DS, Delles C, McClure J, Kingsmore DB. B-type natriuretic peptide predicts postoperative cardiac events and mortality after elective open abdominal aortic aneurysm repair. J Vasc Surg. 2013 Feb;57(2):345-53. doi: 10.1016/j.jvs.2012.07.053. Epub 2012 Oct 9. PMID 23058722
- [Background] Vetrugno L, Costa MG, Pompei L, Chiarandini P, Drigo D, Bassi F, Gonano N, Muzzi R, Della Rocca G. Prognostic power of pre- and postoperative B-type natriuretic peptide levels in patients undergoing abdominal aortic surgery. J Cardiothorac Vasc Anesth. 2012 Aug;26(4):637-42. doi: 10.1053/j.jvca.2012.01.018. Epub 2012 Mar 2. PMID 22387082